CLINICAL TRIAL: NCT06800794
Title: Effect of Meal Timing and Dietary Changes on Metabolic and Behavioral Factors Involved in the Food Insecurity-Obesity Paradox
Brief Title: Investigating Metabolic and Psychological Adaptations in a Clinical Trial
Acronym: IMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008988; 1UM1TR005296-01 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge cluster randomized trial design. Participants are grouped into clusters, which sequentially transition from the control condition to the intervention condition. Each cluster acts as its own control during the baseline period. Data are collected repeatedly over time to evaluate the intervention's effects.
Who Masked: Care Provider
Masking Description: The research assistants who are performing data collection will be blind to what stage of the experiment participants are in. However, the counselor who performs behavioral skills training will not be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): During this phase, participants are told to maintain typical behaviors and not change any normal patterns of activity/eating.
- Treatment phase (Experimental): There are two components to the treatment:
  Food provisioning: The food provisioning component will consist of bi-weekly home deliveries of three meals a day. The number of calories in the provided meals for each day will be personalized based on each participant's resting metabolic rate. Caloric targets for each participant will be 20% of TDEE as this translates to ~1-2 pounds of weight loss per week. Diets composition will also be tailored to help improve TEF and RQ.
  Behavioral Skills Training: This will be based on an evidence-based behavioral weight-loss program developed in our lab. This treatment has shown clinically significant weight loss with positive effects sustained over 10-years. The specific includes lessons on self-monitoring, developing alternatives to foods, meal-planning, goal setting, episodic future thinking, physical activity, and self-reinforcement.
  Interventions: Behavioral: Behavioral Skill Training; Other: Meal Provisioning

INTERVENTIONS:
Behavioral: Behavioral Skill Training — 7 sessions including: Hunger and fullness, eating on a budget, traffic light eating plan, menu planning, creating alternatives to food, financial planning, and changing the environment.
  Arms: Treatment phase
Other: Meal Provisioning — 3 meals a day consisting of low energy dense, nutrient rich, ready to eat, low GI, foods delivered to the participants' homes.
  Arms: Treatment phase

SUMMARY:
This study aims to explore how food insecurity, a lack of consistent access to enough food, may lead to changes in the body that make it harder to lose weight. The investigators are testing whether providing women experiencing food insecurity with a stable, healthy, and personalized meal plan can improve their metabolism and reduce their motivation to eat unhealthy foods. The hypothesis is that addressing food insecurity with a predictable diet can lower a person's respiratory quotient (a measure of how the body uses energy), promote fat burning, and improve overall health. This research will improve the understanding for how food insecurity contributes to obesity and may lead to better solutions for managing weight in individuals facing these challenges.

DETAILED DESCRIPTION:
Women who experience food insecurity have unpredictable access to food and often miss meals and go hungry, but paradoxically are at a 50% greater risk for developing obesity than women who are food secure. This is due in part to metabolic and behavioral factors involved in food insecurity. Research suggests unpredictable access to food is associated with: 1) a high respiratory quotient (RQ) indicative of substrate oxidation that favors storage of fat and burning of carbohydrates; 2) an increase in fuel efficiency and a reduced thermic effect of food (TEF); 3) higher relative reinforcing efficacy of food (RREFOOD), due in part to periodic food deprivation that results from unpredictable access to food and being hungry, and 4) a short temporal window that involves making decisions that focus on meeting immediate versus long-term goals, as assessed by delay discounting (DD). While people with food insecurity and obesity should modify their diet, an RQ that favors storage of fat coupled with a reduced TEF, high RREFOOD and high DD may compromise the effects of traditional dietary approaches to weight loss. The goal of this pilot study is to examine the effects of providing a personalized, stable, predictable, low carbohydrate, low glycemic index, high protein, low energy dense diet on changes in metabolic and behavioral factors that characterize low-income women with food insecurity who have obesity, using a novel stepped wedge design. This work extends our research on behavioral and metabolic factors involved in food insecurity, and will provide strong pilot data for a randomized, controlled trial of a novel dietary approach that target factors involved in food insecurity and obesity that can improve weight control and reduce cardiometabolic risk factors. The investigators expect to screen at least 60 women, with an estimated screen failure rate of 80%. A goal for this pilot project is to provide effect sizes for future studies. The sample size was determined based on feasibility constraints, with the understanding that these results will serve as pilot data for a larger, fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Woman between the ages of 18-45.
* Premenopausal.
* Obese (BMI ≥ 30).
* Diagnosed with prediabetes (HbA1c: 5.7%-6.4%).
* Experiencing food insecurity (score of 2-6 on the six-item food insecurity questionnaire).
* Income below 300% of the household federal poverty threshold.
* Lives alone.

Exclusion Criteria:

* Actively planning to become pregnant (e.g., individuals trying to conceive or undergoing fertility treatment, based on self-report).
* Delivered a baby within the past 6 months (self-report).
* Non-ambulatory (e.g., individuals unable to walk independently or requiring a wheelchair for mobility).
* Intellectual impairment that would impact treatment adherence.
* Unmanaged mood disorders, substance use disorders, personality disorders, or a history of eating disorders, including:

  * Generalized anxiety disorder.
  * Depression.
  * Alcohol dependence.
  * Schizophrenia.
  * Anorexia nervosa, bulimia, or binge eating disorder within the past 6 months.
* Recent weight loss exceeding 5% of body weight within the past 6 months (self-report).
* Food allergies to study-related foods, including dairy, soy, nuts, or gluten.
* History of bariatric surgery or GLP-1 agonist use (self-report).
* Inability to read or write in English (self-report).
* Planned relocation out of the study area during the study timeframe (self-report).
* Uncontrolled diabetes (HbA1c > 9%) or hypertension (blood pressure > 160/100 mmHg), based on self-report or screening visit measurements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Through study completion, an average of 25 weeks
  measured in kgs using a weight scale.
change in HBA1C | Through study completion, an average of 25 weeks.
  measured via a finger-prick blood sample analyzed using a point-of-care device
Change in respiratory quotient | Through study completion, an average of 25 weeks.
  will be measured in morning fasting state using the Breezing Pro, an FDA approved device for portable metabolic measures
change in TEF | Through study completion, an average of 25 weeks.
  will be measured in morning fasting state using the Breezing Pro, an FDA approved device for portable metabolic measures
Change in delay discounting | Through study completion, an average of 25 weeks.
  will be measured using the adjusting amount delay discounting task that presents participants with choices between a fraction of the total delayed amount of money now or the full amount ($100 &/ $1000) at a future delayed time for five different periods from 30 days, 180 days, 365 days (1 year), 1095 days (3 years), 1825 days (5 years) (order randomized).
Change in RRE | Through study completion, an average of 25 weeks.
  RRE will be assessed through a survey that will use participants' preferred snack foods that are classified as either hyperpalatable or healthy. Scores have no fixed minimum or maximum, as they are determined by the highest ratio completed before the participant stops working for the food reward. Higher scores indicate greater reinforcing efficacy and a stronger motivational drive for the food reward, which is considered a worse outcome in this context.

SECONDARY OUTCOMES:
change in stress | Through study completion, an average of 25 weeks.
  measured using the Perceived Stress Scale. The Perceived Stress Scale is a validated 10-item questionnaire that measures the perception of stress over the past month. Scores range from 0 to 40, where higher scores indicate greater perceived stress and worse outcomes.
change in physical activity | Through study completion, an average of 25 weeks.
  measured using a Fitbit activity monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Farber Hall G56, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified individual participant data (IPD) with other researchers to promote transparency, reproducibility, and the advancement of scientific knowledge.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information (Study Protocol, SAP, ICF, and Analytic Code) will be made available no later than 12 months after the publication of the primary study results or 12 months after the final study completion date (November 1, 2025), whichever comes first. Therefore, the anticipated start date for data availability is November 1, 2026. The IPD and supporting information will remain available for a period of 5 years from the start date, allowing sufficient time for secondary analyses and collaborative research. The anticipated end date is November 1, 2031.
Access Criteria: Qualified Researchers: Access will be granted to researchers affiliated with academic, non-profit, or governmental institutions conducting non-commercial research. Researchers must demonstrate a legitimate scientific purpose for using the data.
  Individual Participant Data (IPD):
  De-identified data for all primary and secondary outcome measures (e.g., respiratory quotient, thermic effect of food, body weight, relative reinforcing value of food, and delay discounting).
  Accompanying metadata and codebooks for proper interpretation of the data.
  Supporting Information:
  Study Protocol: Detailed description of the study design and methodology. Statistical Analysis Plan (SAP): Comprehensive explanation of the planned statistical analyses for all outcomes.
  Informed Consent Form (ICF): Template of the consent form used during the study.
  Analytic Code: Scripts used for data cleaning and statistical analyses, enabling reproducibility of results.

REFERENCES:
- [Background] Pannacciulli N, Salbe AD, Ortega E, Venti CA, Bogardus C, Krakoff J. The 24-h carbohydrate oxidation rate in a human respiratory chamber predicts ad libitum food intake. Am J Clin Nutr. 2007 Sep;86(3):625-32. doi: 10.1093/ajcn/86.3.625. PMID 17823426
- [Background] Raynor HA, Epstein LH. The relative-reinforcing value of food under differing levels of food deprivation and restriction. Appetite. 2003 Feb;40(1):15-24. doi: 10.1016/s0195-6663(02)00161-7. PMID 12631501
- [Background] Bickel WK, Freitas-Lemos R, Tomlinson DC, Craft WH, Keith DR, Athamneh LN, Basso JC, Epstein LH. Temporal discounting as a candidate behavioral marker of obesity. Neurosci Biobehav Rev. 2021 Oct;129:307-329. doi: 10.1016/j.neubiorev.2021.07.035. Epub 2021 Aug 3. PMID 34358579
- [Background] Green L, Myerson J, Lichtman D, Rosen S, Fry A. Temporal discounting in choice between delayed rewards: the role of age and income. Psychol Aging. 1996 Mar;11(1):79-84. doi: 10.1037//0882-7974.11.1.79. PMID 8726373
- [Background] Myers CA, Beyl RA, Martin CK, Broyles ST, Katzmarzyk PT. Psychological mechanisms associated with food security status and BMI in adults: a mixed methods study. Public Health Nutr. 2020 Oct;23(14):2501-2511. doi: 10.1017/S1368980020000889. Epub 2020 Jun 29. PMID 32597739
- [Background] Rodriguez LR, Rasmussen EB, Kyne-Rucker D, Wong M, Martin KS. Delay discounting and obesity in food insecure and food secure women. Health Psychol. 2021 Apr;40(4):242-251. doi: 10.1037/hea0001042. PMID 33856831
- [Background] Epstein LH, Truesdale R, Wojcik A, Paluch RA, Raynor HA. Effects of deprivation on hedonics and reinforcing value of food. Physiol Behav. 2003 Feb;78(2):221-7. doi: 10.1016/s0031-9384(02)00978-2. PMID 12576119
- [Background] Crandall AK, Temple JL. Experimental scarcity increases the relative reinforcing value of food in food insecure adults. Appetite. 2018 Sep 1;128:106-115. doi: 10.1016/j.appet.2018.05.148. Epub 2018 May 29. PMID 29852205
- [Background] Myers KP, Majewski M, Schaefer D, Tierney A. Chronic experience with unpredictable food availability promotes food reward, overeating, and weight gain in a novel animal model of food insecurity. Appetite. 2022 Sep 1;176:106120. doi: 10.1016/j.appet.2022.106120. Epub 2022 Jun 6. PMID 35671918
- [Background] Crandall AK, Ziegler AM, Mansouri T, Matteson J, Isenhart E, Carter A, Balantekin KN, Temple JL. Having less and wanting more: an investigation of socioeconomic status and reinforcement pathology. BMC Public Health. 2021 Feb 25;21(1):402. doi: 10.1186/s12889-021-10430-7. PMID 33632174
- [Background] Lin H, Carr KA, Fletcher KD, Epstein LH. Food reinforcement partially mediates the effect of socioeconomic status on body mass index. Obesity (Silver Spring). 2013 Jul;21(7):1307-12. doi: 10.1002/oby.20158. Epub 2013 Jun 11. PMID 23754824
- [Background] Nettle D, Bateson M. Food-Insecure Women Eat a Less Diverse Diet in a More Temporally Variable Way: Evidence from the US National Health and Nutrition Examination Survey, 2013-4. J Obes. 2019 Oct 1;2019:7174058. doi: 10.1155/2019/7174058. eCollection 2019. PMID 31662904
- [Background] Chaput JP, Tremblay A. The glucostatic theory of appetite control and the risk of obesity and diabetes. Int J Obes (Lond). 2009 Jan;33(1):46-53. doi: 10.1038/ijo.2008.221. Epub 2008 Nov 11. PMID 19002144
- [Background] Flatt JP. The difference in the storage capacities for carbohydrate and for fat, and its implications in the regulation of body weight. Ann N Y Acad Sci. 1987;499:104-23. doi: 10.1111/j.1749-6632.1987.tb36202.x. PMID 3300476
- [Background] Ellis AC, Hyatt TC, Hunter GR, Gower BA. Respiratory quotient predicts fat mass gain in premenopausal women. Obesity (Silver Spring). 2010 Dec;18(12):2255-9. doi: 10.1038/oby.2010.96. Epub 2010 May 6. PMID 20448540
- [Background] Booker JM, Chang DC, Stinson EJ, Mitchell CM, Votruba SB, Krakoff J, Gluck ME, Cabeza de Baca T. Food insecurity is associated with higher respiratory quotient and lower glucagon-like peptide 1. Obesity (Silver Spring). 2022 Jun;30(6):1248-1256. doi: 10.1002/oby.23437. PMID 35674698
- [Background] Bateson M, Andrews C, Dunn J, Egger CBCM, Gray F, Mchugh M, Nettle D. Food insecurity increases energetic efficiency, not food consumption: an exploratory study in European starlings. PeerJ. 2021 May 28;9:e11541. doi: 10.7717/peerj.11541. eCollection 2021. PMID 34123601
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Regular meal frequency creates more appropriate insulin sensitivity and lipid profiles compared with irregular meal frequency in healthy lean women. Eur J Clin Nutr. 2004 Jul;58(7):1071-7. doi: 10.1038/sj.ejcn.1601935. PMID 15220950
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Decreased thermic effect of food after an irregular compared with a regular meal pattern in healthy lean women. Int J Obes Relat Metab Disord. 2004 May;28(5):653-60. doi: 10.1038/sj.ijo.0802616. PMID 15085170
- [Background] Calcagno M, Kahleova H, Alwarith J, Burgess NN, Flores RA, Busta ML, Barnard ND. The Thermic Effect of Food: A Review. J Am Coll Nutr. 2019 Aug;38(6):547-551. doi: 10.1080/07315724.2018.1552544. Epub 2019 Apr 25. PMID 31021710
- [Background] Morales ME, Berkowitz SA. The Relationship between Food Insecurity, Dietary Patterns, and Obesity. Curr Nutr Rep. 2016 Mar;5(1):54-60. doi: 10.1007/s13668-016-0153-y. Epub 2016 Jan 25. PMID 29955440
- [Background] Franklin B, Jones A, Love D, Puckett S, Macklin J, White-Means S. Exploring mediators of food insecurity and obesity: a review of recent literature. J Community Health. 2012 Feb;37(1):253-64. doi: 10.1007/s10900-011-9420-4. PMID 21644024
- [Background] Nettle D, Andrews C, Bateson M. Food insecurity as a driver of obesity in humans: The insurance hypothesis. Behav Brain Sci. 2017 Jan;40:e105. doi: 10.1017/S0140525X16000947. Epub 2016 Jul 28. PMID 27464638
- [Background] Bateson M, Pepper GV. Food insecurity as a cause of adiposity: evolutionary and mechanistic hypotheses. Philos Trans R Soc Lond B Biol Sci. 2023 Oct 23;378(1888):20220228. doi: 10.1098/rstb.2022.0228. Epub 2023 Sep 4. PMID 37661744
- [Background] Epstein LH, Rizwan A, Paluch RA, Temple JL. Delay Discounting and the Income-Food Insecurity-Obesity Paradox in Mothers. J Obes. 2023 Sep 19;2023:8898498. doi: 10.1155/2023/8898498. eCollection 2023. PMID 37766882
- [Background] Epstein LH, Jankowiak N, Lin H, Paluch R, Koffarnus MN, Bickel WK. No food for thought: moderating effects of delay discounting and future time perspective on the relation between income and food insecurity. Am J Clin Nutr. 2014 Sep;100(3):884-90. doi: 10.3945/ajcn.113.079772. Epub 2014 Jul 9. PMID 25008855